CLINICAL TRIAL: NCT02511236
Title: Addressing Racial/Ethnic Tobacco Health Disparities Via Group Intervention
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: H. Lee Moffitt Cancer Center and Research Institute (Other); James and Esther King Biomedical Research Program (Other)
Responsible Party: Principal Investigator, David Lee, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20150356
Record Dates: First submitted 2015-07-24; First posted 2015-07-29 (Estimated); Results first posted 2021-06-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group Cognitive Behavioral Therapy (Experimental): Participants may receive 8 group cognitive behavioral therapy (CBT) sessions and eight weeks of transdermal nicotine patches (TNP) [21mg (4 weeks), 14mg (2 weeks), and 7mg (2 weeks)].
  Interventions: Behavioral: Group Cognitive Behavioral Therapy; Drug: Transdermal Nicotine Patch
- General Health Education (Active Comparator): Participants may receive group general health education (GHE) sessions and eight weeks of transdermal nicotine patches (TNP) [21mg (4 weeks), 14mg (2 weeks), and 7mg (2 weeks)].
  Interventions: Behavioral: General Health Education; Drug: Transdermal Nicotine Patch

INTERVENTIONS:
Behavioral: Group Cognitive Behavioral Therapy — The four-week CBT protocol includes 4 sessions during week 1, 2 sessions during week 2, 1 session during week 3, and 1 session during week 4. Sessions may include a functional analysis of smoking patterns, environmental cues, and motivation for change, and cover nicotine addiction and withdrawal, health consequences, benefits of cessation, stress management, negative affect, alcohol use, triggers, coping responses, cognitive restructuring, social support, decision making, weight control, and physical activity.
  Arms: Group Cognitive Behavioral Therapy
Behavioral: General Health Education — The four-week CBT protocol includes 4 sessions during week 1, 2 sessions during week 2, 1 session during week 3, and 1 session during week 4. Sessions may include didactic information on tobacco-associated morbidities, such as heart disease, diabetes, and hypertension. Content may include Power Point-delivered lectures on the prevalence, etiology, basic pathology, symptom patterns, and treatment of the conditions, and discussion questions designed to facilitate learning and interest. Smoking cessation specific topics will not be addressed, and coping skills will not be provided. Participants will be allowed to share feelings regarding smoking (if they mention them) and general questions will be answered, although no specific behavioral quitting advice will be provided (i.e., they will be encouraged to adhere to the TNP protocol).
  Arms: General Health Education
Drug: Transdermal Nicotine Patch — Participants will be prescribed up to 8 weeks of transdermal nicotine patch therapy, including 21 mg for 4 weeks, 14 mg for 2 weeks, and 7 mg for 2 weeks. Dosages will be adjusted per manufacturer recommendations.
  Other Names: Nicotine Patch

SUMMARY:
The purpose of this study is to test the effects of a group smoking cessation program. The study will also examine individual differences in response to the intervention program.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as African American/Black, Hispanic (any race), or White non-Hispanic
* Smoke at least 5 cigarettes/day or carbon monoxide (CO) reading of at least 8 ppm
* be over age 18
* speak/read English and/or Spanish

Exclusion Criteria:

* Contraindications for transdermal nicotine patch therapy (TNP)
* Cognitive or mental health impairment that inhibits group treatment
* Currently being treated for smoking cessation, alcoholism, or illicit drug use
* Unable to attend sessions
* Indications that participant is not appropriate for the study (e.g., aggressive, intoxicated, disruptive, visibly ill)
* Does not self-identify as African American, Hispanic, or White (non-Hispanic)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2015-08; Primary Completion 2019-10-23 (Actual); Study Completion 2019-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Lee, PhD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - University of Miami, Coral Gables, Florida
  - H Lee Moffitt Cancer Center, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Webb Hooper M, Lee DJ, Simmons VN, Brandon KO, Antoni MH, Asfar T, Koru-Sengul T, Brandon TH. Cognitive behavioral therapy versus general health education for smoking cessation: A randomized controlled trial among diverse treatment seekers. Psychol Addict Behav. 2024 Feb;38(1):124-133. doi: 10.1037/adb0000928. Epub 2023 May 4. PMID 37141036
- [Derived] Webb Hooper M, Lee DJ, Simmons VN, Brandon KO, Antoni MH, Unrod M, Asfar T, Correa JB, Koru-Sengul T, Brandon TH. Reducing racial/ethnic tobacco cessation disparities via cognitive behavioral therapy: Design of a dualsite randomized controlled trial. Contemp Clin Trials. 2018 May;68:127-132. doi: 10.1016/j.cct.2018.03.017. Epub 2018 Apr 1. PMID 29617633

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group Cognitive Behavioral Therapy | General Health Education
Started | 165 | 191
Completed | 125 | 146
Not Completed | 40 | 45

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group Cognitive Behavioral Therapy | General Health Education | Total
Number analyzed (Participants) | 165 | 191 | 356
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.13 (10.73) | 51.86 (10.71) | 51.08 (10.73)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 83 | 97 | 180
  Male | 81 | 94 | 175
  Unknown | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 47 | 137 | 184
  Not Hispanic or Latino | 116 | 52 | 168
  Unknown or Not Reported | 2 | 2 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 78 | 81 | 159
  Black/African American | 63 | 81 | 144
  Native American | 0 | 2 | 2
  Other | 24 | 27 | 51
Total Household Income [Number; unit: participants]
  Under $10,000 | 49 | 73 | 122
  $10,000-$20,000 | 36 | 36 | 72
  $20,001-$30,000 | 21 | 20 | 41
  $30,001-$40,000 | 15 | 10 | 25
  $40,001-$50,000 | 10 | 11 | 21
  $50,001-$60,000 | 10 | 13 | 21
  $60,001-$70,000 | 7 | 4 | 11
  $70,001-$80,000 | 2 | 3 | 5
  $80,001-$90,000 | 3 | 4 | 7
  Over $90,000 | 9 | 14 | 23
  Unknown | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Reporting 7 Day Point Prevalence Abstinence
Description: Reported will be the number of participants reporting 7 day point prevalence of smoking abstinence
Time Frame: 12-months
Population: Not all participants that completed the 12 month follow up visit were able to report their 7 day point prevalence abstinence
Measure: Count of Participants; unit: Participants
Arm/Group | Group Cognitive Behavioral Therapy | General Health Education
Number analyzed (Participants) | 97 | 113
Participants | 54 | 45

2. Primary Outcome: Change in Perceived Stress Scores
Description: The Perceived Stress Scale (PSS) is a 10-item questionnaire with scores ranging from 0-40 with higher scores indicated greater stress.
Time Frame: Baseline, 4 weeks
Population: Not all participants that completed the 4 week follow up visit were able to complete the PSS questionnaire
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Group Cognitive Behavioral Therapy | General Health Education
Number analyzed (Participants) | 118 | 139
score on a scale | -1.47 (0.502) | -1.85 (0.534)

3. Primary Outcome: Change in Depressive Symptoms Scores
Description: Depressive scores based on Center for Epidemiologic Studies Depression Scale (CESD). CESD has a total score ranging from 0-60 with a higher score indicating greater depressive symptoms.
Time Frame: Baseline, 4 weeks
Population: Not all participants that completed the 4 week follow up visit were able to complete the CESD questionnaire
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Group Cognitive Behavioral Therapy | General Health Education
Number analyzed (Participants) | 116 | 140
score on a scale | -1.84 (0.841) | -1.53 (0.803)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Group Cognitive Behavioral Therapy | General Health Education
All-Cause Mortality (participants affected / at risk) | 0/165 | 4/191
Serious Adverse Events (participants affected / at risk) | 0/165 | 4/191
Other Adverse Events (participants affected / at risk) | 2/165 | 0/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group Cognitive Behavioral Therapy (N=165) | General Health Education (N=191)
Death/Suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1)
Death (Immune system disorders) | 0 (0) | 1 (1)
Death (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group Cognitive Behavioral Therapy (N=165) | General Health Education (N=191)
Achillese tendon injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-11): https://cdn.clinicaltrials.gov/large-docs/36/NCT02511236/Prot_SAP_000.pdf